CLINICAL TRIAL: NCT01062100
Title: The Hamilton Prospective Pilot Study To Investigate the Feasibility and Safety of A Dedicated High Resolution Nuclear Breast Imaging Camera
Brief Title: Study To Investigate the Feasibility and Safety of A Dedicated High Resolution Nuclear Breast Imaging Camera
Acronym: THORN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCOG-2009-THORN
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; molecular breast imaging; MRI; gamma camera
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nuclear breast imaging (Experimental): nuclear breast imaging using MBI Gamma camera
  Interventions: Device: nuclear breast imaging using MBI Gamma camera

INTERVENTIONS:
Device: nuclear breast imaging using MBI Gamma camera — nuclear breast imaging using MBI Gamma camera in addition to MRI

SUMMARY:
To evaluate the feasibility, acceptability and safety of using a molecular breast imaging (MBI) Gamma Camera in women at high risk of developing breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Females ≥18 years of age
* Undergoing annual breast MRI because of a high risk of breast cancer due to any of the following:

  * Known BRCA1 or BRCA2 mutation carriers, or is untested for BRCA but is a first degree relative of a BRCA mutation carrier
  * History of radiation to the chest between 10-30 years of age (e.g. Hodgkin's Disease)
  * History of Cowdens or Li Fraumeni Syndrome
  * A first degree relative with Cowdens or Li Fraumeni Syndrome
  * Prior breast biopsy positive for lobular carcinoma in situ (LCIS) or atypical lobular hyperplasia or atypical ductal hyperplasia (ADH)
  * Family history consistent with a hereditary breast cancer syndrome and estimated personal lifetime cancer risk ≥25% using the IBIS risk evaluator

Exclusion Criteria:

* Pregnant or lactating
* History of invasive breast cancer or ductal carcinoma in situ (DCIS)
* Unable to undergo MRI because of:

  * Renal dysfunction with an estimated creatinine clearance of < 30 ml/min calculated using the Cockcroft-Gault formula
  * Implanted ferrous metal prostheses
  * Claustrophobia
  * Medical or psychological conditions that on assessment, make them unable to complete the procedure
  * Known allergies to Gadolinium-DTPA
* Known allergies to Sestamibi (Miraluma or Cardiolite)
* Prior bilateral mastectomy
* Prior breast biopsy or surgery within 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility, safety and acceptability to patients of the MBI Gamma camera. | 1 year

SECONDARY OUTCOMES:
To explore the ability of the MBI Gamma camera to detect breast cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Pond, Principal Investigator — Ontario Clinical Oncology Group - McMaster University; Karen Gulenchyn, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada